CLINICAL TRIAL: NCT03454490
Title: Pseudoaneurysm of the Greater Palatine Artery Following Autogenous Connective Tissue Gingival Graft : A Case Series
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hopital de l'Enfant-Jesus (Other)
Responsible Party: Principal Investigator, Simon Jean, Principal Investigator, Hopital de l'Enfant-Jesus
Other Study IDs: Postoperative pseudoaneurysm
Record Dates: First submitted 2018-02-22; First posted 2018-03-06 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Pseudoaneurysm
Keywords: Gingival graft; Pseudoaneurysm; Postoperative complication; Gingival recession treatment; Palatine mass; Palatine bleeding
MeSH Terms: conditions — Aneurysm, False; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Postoperative pseudoaneurysm of the greater palatine artery — Patients had an autogenous connective tissue gingival graft.

SUMMARY:
Gingival recession is defined as the apical migration of the gingival margin from the amelocemental junction. This condition may be associated with symptoms such as tooth hypersensitivity, root decay, and cosmetic complaints from patients. Many treatments have been used to treat gingival recession and the gold standard is the autogenous connective tissue gingival graft because of its predictability. This type of gingival graft is performed by harvesting connective tissue from patients' hard palate. Periodontists and general dentists frequently perform these gingival grafts. Occasionally, some patients develop postoperative complications that need to be addressed in an hospital setting. An uncommon but concerning complication of an autogenous connective tissue gingival graft is a donor site pseudoaneurysm of the greater palatine artery. No description of this complication following a gingival graft has been identified in the current literature. One case report mentioned that pseudoaneurysm of the greater palatine artery looks like a pulsatile nodule associated or not with pain on palpation. From the experience of the investigators, patients may consult an hospital setting having a complaint of major oral bleeding. Local hemostatic agents can palliate this type of bleeding, but angiographic embolization is often required. Several cases were treated in the investigators' hospital. Thus, the investigators believe it is relevant to share this experience with the scientific community. The primary objective of this case series is to inform dental professionals of the existence and the management of postoperative pseudoaneurysm of the greater palatine artery following autogenous gingival graft. The secondary objective is to find potential solutions to minimize the incidence of this morbid complication.

ELIGIBILITY:
Inclusion Criteria:

* Population : Patients having a diagnostic of pseudoaneurysm of the greater palatine artery who had an autogenous connective tissue gingival graft
* Intervention : Patients treated with local hemostatic agents or by angiographic embolization
* Comparison : None

Exclusion Criteria:

* Missing data in patients' chart precluding complete data extraction

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients having a diagnostic of pseudoaneurysm of the greater palatine artery who had an autogenous connective tissue gingival graft
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative oral bleeding | One month following autogenous connective tissue gingival graft
  Complication following autogenous connective tissue gingival graft

SECONDARY OUTCOMES:
Use of local hemostatic agents | Six months
  Palliative method before definitive care
Secondary effects following angiographic intervention | Six months
  Postoperative infection, bone or gum necrosis, extrusion of embolization material, loss of tooth, tooth devitalization following angiographic intervention
Number of followups required | Six months
  Secondary effects following angiographic intervention

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Paris, DMD, FRCD, Study Director — Hopital de l'Enfant-Jesus, CHU de Quebec, Laval University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yadav AP, Kulloli A, Shetty S, Ligade SS, Martande SS, Gholkar MJ. Sub-epithelial connective tissue graft for the management of Miller's class I and class II isolated gingival recession defect: A systematic review of the factors influencing the outcome. J Investig Clin Dent. 2018 Aug;9(3):e12325. doi: 10.1111/jicd.12325. Epub 2018 Feb 9. PMID 29424485
- [Background] Tozum TF, Keceli HG, Guncu GN, Hatipoglu H, Sengun D. Treatment of gingival recession: comparison of two techniques of subepithelial connective tissue graft. J Periodontol. 2005 Nov;76(11):1842-8. doi: 10.1902/jop.2005.76.11.1842. PMID 16274302
- [Background] Byun HY, Oh TJ, Abuhussein HM, Yamashita J, Soehren SE, Wang HL. Significance of the epithelial collar on the subepithelial connective tissue graft. J Periodontol. 2009 Jun;80(6):924-32. doi: 10.1902/jop.2009.080673. PMID 19485822
- [Background] Thomas J, Patel NS, Viroslav A, Sheykholeslami K. Greater palatine artery pseudoaneurysm presenting as a slow-growing palatal mass. J Oral Maxillofac Surg. 2013 Apr;71(4):e164-7. doi: 10.1016/j.joms.2012.11.017. Epub 2013 Jan 29. No abstract available. PMID 23375075